CLINICAL TRIAL: NCT00626652
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Dose-escalation Study of the Effects of K201 Injection, 2 mg/mL on the Restoration of Sinus Rhythm in Subjects Who Are in Atrial Fibrillation
Brief Title: Study of K201 Injection on Restoration of Sinus Rhythm in Subjects Who Are in Atrial Fibrillation
Acronym: RESTORATION
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sequel Pharmaceuticals, Inc (Industry)
Responsible Party: Howard C. Dittrich, MD; Chief Medical Officer, Sequel Pharmaceuticals
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CJI-201
Record Dates: First submitted 2008-02-18; First posted 2008-02-29 (Estimated); Last update posted 2010-01-08 (Estimated); Status verified 2010-01

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — K201 compound

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: K201 Injection

INTERVENTIONS:
Drug: K201 Injection — single intravenous infusion of Dose 1 - 10 or placebo (saline) or single oral capsule Dose A or placebo capsule

SUMMARY:
To evaluate the effects of K201 on sinus rhythm restoration, symptom score, various cardiovascular parameters, and safety.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic atrial fibrillation
* Atrial fibrillation documented by ECG
* Adherence to local clinical standards or the ACC/AHA/ESC practice guidelines for atrial fibrillation regarding thrombo-embolic event prevention and treatment.

Exclusion Criteria:

* Systolic blood pressure <100 mmHg
* Heart rate <50 bpm
* Temperature >38°C
* QT or QTcB >440 ms
* QRS >140 ms
* Paced atrial or ventricular rhythm on ECG
* Serum potassium <3.5 meq/L
* History of receiving another intravenous Class I or Class III antiarrhythmic drug within 3 days of randomization
* History of amiodarone in last 6 months.
* Clinical evidence of acute coronary syndrome
* Acute pulmonary edema or embolism
* Hyperthyroidism
* Acute pericarditis
* History of failed electrical cardioversion at any time
* History of torsades des pointes
* History of familial long QT interval syndrome
* History of ventricular tachycardia requiring drug or device therapy
* History of NYHA Heart Failure Class 3 or 4.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2008-03; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Restoration of sinus rhythm | 24hrs

CONTACTS AND LOCATIONS:
Overall Officials: Sergey Pavlovich Golitsyn, Prof., Principal Investigator — Russian Cardiologic Scientific and Manufacturing Complex of Roszdrav, Institute of Cardiology n.a. A.L.Myasnikov, Department of clinical electrophysiology; Amos Katz, Prof., Principal Investigator — Barzilai Medical Center
Locations (9):
- Israel (7):
  - Ashkelon
  - Beersheba
  - Haifa
  - Holon
  - Jerusalem
  - Nazareth
  - Safed
- Russia (2):
  - Moscow
  - Saint Petersburg